CLINICAL TRIAL: NCT06735261
Title: Evaluation of the Efficacy of Sphenopalatine Block in Headache in Patients With Non-traumatic Subarachnoid Hemorrhage (SAH) After Training of Neurosurgical Intensive Care Nurses.
Brief Title: Sphenopalatine Block in Headache in Patients With Non-traumatic Subarachnoid Hemorrhage
Acronym: SATURN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHU GRENOBLE ALPES / SATURN
Record Dates: First submitted 2024-12-03; First posted 2024-12-16 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Subarachnoid Hemorrhage in Adult Patients
Keywords: pain; adulte; intensive care; subarachnoid hemorrhage; securing aneurysm; lidocaine
MeSH Terms: conditions — Pain; Subarachnoid Hemorrhage | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, randomized, open-label study,
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Pain management according to the protocol in force in the neurosurgical intensive care unit (analgesics: Paracetamol, Nefopam and morphine PCA).
- Sphenopalatine Ganglion Block using 2% lidocaine (Experimental): Addition of (BGSP) Sphenopalatine ganglion block with Lidocaine 2% Injectable Solution (2mg/ml) 1.5ml * 3 consecutive times maximum if EN >3/10, to be repeated every 12h for 7 days if necessary. BGSP performed by the department's Ides after training by the anesthetists.

INTERVENTIONS:
Procedure: Sphenopalatine Ganglion Block using 2% lidocaine — A hollow-stem swab soaked in viscous Xylocaine is inserted into the patient's nasal cavity (one swab per nostril) until it stops. 1.5ml Lidocaine 20% (20mg/ml) is injected into each swab using a 5ml syringe and a pink trocar. Both swabs are left in place for 10 min.

SUMMARY:
Non-traumatic SAH, linked in 85% of cases to the rupture of an intracranial aneurysm, is a serious stroke affecting young people. Half of all survivors suffer cognitive impairment. The presentation is that of a sudden-onset, isolated headache. This population is exposed to headache during hospitalization, which lasts an average of 13 days. This length of hospitalization is due to the fact that these patients must be monitored during the potential vasospasm period that occurs between days 4 and 14 after SAH. The pain associated with SAH is a source of discomfort and increased morphine consumption during the ICU stay, particularly during the first 10 days. Current recommendations call for conventional pain management with a combination of tier 1, 2 and/or 3 analgesics. For headache control, opioids are widely prescribed, sometimes in high doses, with adverse effects, despite efforts to reduce their use. Maximum headache pain scores remain high, indicating inadequate pain management. This highlights the urgent need to study alternative opioid-sparing and analgesia strategies for patients with SAH.

DETAILED DESCRIPTION:
Sphenopalatine block is already used for certain types of facial and cranial pain, and could help save morphine consumption during hospitalization. The sphenopalatine ganglion is a crossroads for parasympathetic, sympathetic and sensory pathways. Recently studied in post-puncture dural breaches with promising results, sphenopalatine ganglion block (SPGN) may appear as an interesting alternative therapy in the treatment of SAH headaches. Other advantages of this block are its simplicity, efficacy and the absence of any noticeable adverse effects at the time it is performed. What's more, it is already used routinely in our department, with rapid and effective action. The hypothesis of the trial would be to reduce morphine consumption by at least 50% for patients benefiting from BGSP, for better neurological monitoring and optimal overall pain management in SAH.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Non-traumatic SAH with or without aneurysm on brain imaging
* WFNS score 1 and 2
* Patient awake and extubated after radiological procedure
* Patient in pain (EN > 3/10) despite usual level 1 analgesics (Paracetamol + Acupan)
* Affiliated with or benefiting from a social security scheme

Exclusion Criteria:

* Contraindication to sphenopalatine ganglion block (deviated nasal septum, repeated epistaxis, allergy to Lidocaine)
* Patient unable to assess pain by EN
* Persons covered by Articles L1121-5 to L1121-8 of the CSP and Articles 31 to 35 of Regulation 536/2014.
* Participation in other interventional research
* Patient's refusal to participate
* Arteriography more than 48 hours old
* Inaugural headache lasting more than 48 hours
* Presence of an unsecured vascular malformation at high risk of rupture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Demonstrate a 50% change in morphine consumption with sphenopalatine ganglion block during the first 72 hours after cerebral arteriography | during 72 hours
  Total morphine consumption in mg in the first 72 hours after cerebral arteriography in the Intensive care (ICU)

SECONDARY OUTCOMES:
Demonstrate a significant 3-point change in pain on EN (Simple Numerical Scale)averaged over 7 days after arteriography | during 7 days
  EN (Simple Numerical Scale) 7-day average
Describe morphine consumption per day during the patient's hospitalization for the 2 groups | during hospitalization or 10 days
  Morphine consumption in mg per day during hospitalization.
Describe the complications associated with sphenopalatine ganglion block. | during 7 days
  Complications of the sphenopalatine ganglion block technique: incidence of soft palate anesthesia (false liquid routes at H+2), epistaxis, vasovagal reactions, transient hearing loss
Evaluate the feasibility of the (BGSP) sphenopalatine ganglion block act performed by Ides | during 7 days
  Number of sphenopalatine ganglion block (BGSP) failures
Demonstrate that the sphenopalatine ganglion block strategy changes headaches at 28 days. | at 28 days
  EN (Simple Numerical Scale) at Day 28, consumption of stage 3 analgesics or neuropathic
Demonstrate that the sphenopalatine ganglion block strategy changes patient satisfaction at Day 28 | at 28 days
  Questionnaire on overall satisfaction with pain management
Evaluation of nursing practices on the BGSP technique | up to 28 days
  Satisfaction questionnaire for nurses

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nair AS, Rayani BK. Sphenopalatine ganglion block for relieving postdural puncture headache: technique and mechanism of action of block with a narrative review of efficacy. Korean J Pain. 2017 Apr;30(2):93-97. doi: 10.3344/kjp.2017.30.2.93. Epub 2017 Mar 31. PMID 28416992
- [Background] Hung KC, Chen JY, Ho CN, Sun CK. Use of sphenopalatine ganglion block in patients with postdural puncture headache: a pilot meta-analysis. Br J Anaesth. 2021 Jan;126(1):e25-e27. doi: 10.1016/j.bja.2020.10.005. Epub 2020 Oct 31. No abstract available. PMID 33131755
- [Background] Cohen S, Levin D, Mellender S, Zhao R, Patel P, Grubb W, Kiss G. Topical Sphenopalatine Ganglion Block Compared With Epidural Blood Patch for Postdural Puncture Headache Management in Postpartum Patients: A Retrospective Review. Reg Anesth Pain Med. 2018 Nov;43(8):880-884. doi: 10.1097/AAP.0000000000000840. PMID 30063655
- [Background] Viswanathan V, Lucke-Wold B, Jones C, Aiello G, Li Y, Ayala A, Fox WC, Maciel CB, Busl KM. Change in opioid and analgesic use for headaches after aneurysmal subarachnoid hemorrhage over time. Neurochirurgie. 2021 Sep;67(5):427-432. doi: 10.1016/j.neuchi.2021.03.006. Epub 2021 Mar 23. PMID 33771620
- [Background] Kent S, Mehaffey G. Transnasal sphenopalatine ganglion block for the treatment of postdural puncture headache in obstetric patients. J Clin Anesth. 2016 Nov;34:194-6. doi: 10.1016/j.jclinane.2016.04.009. Epub 2016 May 11. PMID 27687372
- [Background] Takmaz SA, Karaoglan M, Baltaci B, Bektas M, Basar H. Transnasal Sphenopalatine Ganglion Block for Management of Postdural Puncture Headache in Non-Obstetric Patients. J Nippon Med Sch. 2021;88(4):291-295. doi: 10.1272/jnms.JNMS.2021_88-406. PMID 34471063
- [Background] Siegler BH, Dos Santos Pereira RP, Kessler J, Wallwiener S, Wallwiener M, Larmann J, Picardi S, Carr R, Weigand MA, Oehler B. Intranasal Lidocaine Administration via Mucosal Atomization Device: A Simple and Successful Treatment for Postdural Puncture Headache in Obstetric Patients. Biomedicines. 2023 Dec 13;11(12):3296. doi: 10.3390/biomedicines11123296. PMID 38137518
- [Background] Singh S, Iqbal J, Jahan N, Yadav R. Sphenopalatine Ganglion Block for the Treatment of Severe Headache following a Ruptured Aneurysm. Neurol India. 2022 Nov-Dec;70(6):2452-2453. doi: 10.4103/0028-3886.364060. No abstract available. PMID 36537435
- See also: Lidocaine Toxicity — https://www.ncbi.nlm.nih.gov/books/NBK482479/